CLINICAL TRIAL: NCT03177096
Title: Impact of the Continuous Measurement of Blood Glucose on Insulin Pump on Child Quality of Life With Type 1 Diabetes. A French Monocentric Prospective Study (IM-CAPT)
Brief Title: Impact of the Continuous Measurement of Blood Glucose on Insulin Pump on Child Quality of Life With Type 1 Diabetes
Acronym: IM-CAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GHR 866; 2016-A01264-47 (Other: Agence Nationale Sécurité du Médicament et produits de santé)
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2018-05

CONDITIONS: Type1diabetes
Keywords: Type 1 diabetes children,School,Childcare facilities,Sensor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peds QL questionnaire and diabetes modulate (Experimental): Routine practice of a continuous measure sensor of the glycemia with insulin pump for children aged 2 to 13 years followed at Mulhouse Hospital for type 1 diabetes : 5 sessions after enrollment visit(V1) (1 session 2 months, 4 months, 6 months, 8 months and 10 months) This study will be proposed to patients treated for type 1 diabetes enrolled in kindergarten, primary school, attending a nursery or a childcare center (patient's participation = 10 months) and will evaluate the child quality of life and the parents and staffs in preschool and school felt too.
  Interventions: Behavioral: Peds QL questionnaire and diabetes modulate; Behavioral: WHO-5 questionnaire; Behavioral: Felt questionnaire

INTERVENTIONS:
Behavioral: Peds QL questionnaire and diabetes modulate — Peds QL questionnaire and diabetes modulate is a pediatric questionnaire about quality of life - children's version and parents version : assessed in the 1st visit (enrollment visit) and after ten months ( V6 End of study)
Behavioral: WHO-5 questionnaire — WHO-5 questionnaire is a questionnaire about quality of life : assessed in the 1st visit (enrollment visit) and after ten months (V6 End of Study) by the children
Behavioral: Felt questionnaire — Felt questionnaire completed by parents with regard to the welcome of their child in community and by the staffs in preschool, school or in out-of school center : assessed 2 months (V2) and ten months (V6 End of study) after enrollment visit

SUMMARY:
The implementation of a sensor of glycemia Enlite coupled with an insulin pump (Medtronic Minimed 640G) is a therapeutic option that Hospital of Mulhouse can propose to the children affected by type 1 diabetes. The glycemic rate detected by the sensor of continuous measure of the glycemia is visible in real time on the pump and then the rate can be normalized. The study will evaluate the impact of the continuous measurement of blood glucose on insulin pump on child quality of life with type 1 diabetes aged 2 to 13 years old.

DETAILED DESCRIPTION:
The French High Health Authority recommends, for patient with type1 diabetes, a supervision of at least 4 tests a day in pre and post prandial with additional controls in circumstances of meal or of unusual physical activities.

Du to age, this control need supervision of an adult, in each place of children life (school, nursery, out-of-school center ...), according to their autonomy.

During several years, all the actors of educational care tried to improve the welcome of the children affected by handicap or by chronic disease.

Since 10 years, the team of pediatric diabetology of Mulhouse Hospital has developed a partnership with the department of Education by setting up every year in September of a training courses for voluntary teachers and all staff nursery.

These sessions are consisted of a formal time bringing knowledge on the disease, followed by exchanges and finally a practical time around manipulation of the readers of glycemia and pumps.

Alerts can be scheduled to warm an increase or an important reduction of blood glucose.

The study will evaluate the child quality of life, and also parents and staffs in preschool, school or in out-of-school center felt too.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment between September 15 to November 15, 2016
* Insulin-dependent Type 1 Diabetes with insulin pump
* From 2 to 13 years old
* Schooled to the nursery or primary school, seeing frequently a day-nursery or in an out-of-school center
* Treated at the hospital of Mulhouse, France

Exclusion Criteria:

* Opposition to study participation
* Patients who don't need sensor of measure of the continuous glycemia

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Evolution of Peds QL questionnaire results | Through study completion, an average of 10 months
  Questionnaire of quality of life (QL)

SECONDARY OUTCOMES:
Evolution of WHO-5 and felt questionnaire | through study completion, an average of 10 months
  Questionnaire of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Fatiha GUEMAZI-KHEFFI, MD, Principal Investigator
Locations (1):
- GHRMSA, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rewers MJ, Pillay K, de Beaufort C, Craig ME, Hanas R, Acerini CL, Maahs DM; International Society for Pediatric and Adolescent Diabetes. ISPAD Clinical Practice Consensus Guidelines 2014. Assessment and monitoring of glycemic control in children and adolescents with diabetes. Pediatr Diabetes. 2014 Sep;15 Suppl 20:102-14. doi: 10.1111/pedi.12190. No abstract available. PMID 25182311
- [Background] Danne T, Tsioli C, Kordonouri O, Blaesig S, Remus K, Roy A, Keenan B, Lee SW, Kaufman FR. The PILGRIM study: in silico modeling of a predictive low glucose management system and feasibility in youth with type 1 diabetes during exercise. Diabetes Technol Ther. 2014 Jun;16(6):338-47. doi: 10.1089/dia.2013.0327. Epub 2014 Jan 21. PMID 24447074
- [Background] Conget I, Choudhary P, Olsen BS et al. Prevention of hypoglycaemia by the predictive low glucose management feature in a user evaluation study. abstract #865
- [Background] Choudhary P, Olsen BS, Conget I, Welsh JB, Vorrink L, Shin JJ. Hypoglycemia Prevention and User Acceptance of an Insulin Pump System with Predictive Low Glucose Management. Diabetes Technol Ther. 2016 May;18(5):288-91. doi: 10.1089/dia.2015.0324. Epub 2016 Feb 23. PMID 26907513
- [Background] Besbes H, Hammami S et al. SFP P-024 - Etude de la qualité de vie des enfants atteints de diabète de type 1 ; Archives de Pédiatrie Volume 21, Issue 5, Supplement 1, May 2014, Pages 734
- [Background] Varni JW, Burwinkle TM, Jacobs JR, Gottschalk M, Kaufman F, Jones KL. The PedsQL in type 1 and type 2 diabetes: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales and type 1 Diabetes Module. Diabetes Care. 2003 Mar;26(3):631-7. doi: 10.2337/diacare.26.3.631. PMID 12610013
- [Background] Institut de Veille Sanitaire. Prévalence et incidence du diabète / Données épidémiologiques / Diabète / Maladies chroniques et traumatismes / Dossiers thématiques / Accueil